CLINICAL TRIAL: NCT04446715
Title: Comparison of Clinical Effects of Meperidine and Sufentanil Added to 0.5% Hyperbaric Bupivacaine for Spinal Anesthesia in Patients Undergoing Cesarean Section
Brief Title: Comparison of Meperidine and Sufentanil Added to 0.5% Hyperbaric Bupivacaine for Spinal Anesthesia in Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Saleh Kanawati, Acting chairperson, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 17062020
Record Dates: First submitted 2020-06-19; First posted 2020-06-25 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Sufentanil; Meperidine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sufentanil Group (Experimental): Patients will receive sufentanil 5 μg in addition to 0.5% heavy bupivacaine spinal anesthesia
  Interventions: Drug: sufentanil; Drug: Bupivacaine
- Meperidine Group (Experimental): Patients will receive meperidine 12.5 mg in addition to 0.5% heavy bupivacaine spinal anesthesia
  Interventions: Drug: meperidine; Drug: Bupivacaine

INTERVENTIONS:
Drug: sufentanil — Patients will receive sufentanil in spinal anesthesia
  Arms: Sufentanil Group
Drug: meperidine — Patients will receive meperidine in spinal anesthesia
  Arms: Meperidine Group
Drug: Bupivacaine — Patients will receive 0.5% heavy bupivacaine in spinal anesthesia

SUMMARY:
Subarachnoid block is a widely used anesthetic technique for cesarean section. To improve the quality of analgesia and prolong its duration, the addition of intrathecal opioids to local anesthetics has been encouraged.

In a double blind randomized controlled trial, 60 parturient women ASA 2-3 scheduled for elective cesarean delivery under spinal anesthesia will be randomly divided into 2 groups: Group 1 will receive sufentanil 5 μg and Group 2 will receive meperidine 12.5 mg. In every group, 0.5% heavy bupivacaine 10 will be added.

DETAILED DESCRIPTION:
A questionnaire will be used to collect data. Patients' demographic and operative characteristics will be recorded. These include block level, heart rate, mean arterial pressure, nausea, vomiting, shivering and use of vasopressors. Post-operative data include pain, analgesic consumption, nausea and vomiting, as well as patients and surgeons satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women with American Society of Anesthesiologist (ASA) 2-3
* scheduled for elective cesarean section.

Exclusion Criteria:

* refuse to participate in the study,
* requiring emergency obstetric care,
* ASA IV or V,
* having systemic diseases,
* a known fetal anomaly,
* placenta previa,
* abruption placenta
* with a history of hypersensitivity or allergy to any of the study drugs,
* operation time longer than 1.5 hour,
* blood loss more than 1500 millilitres,
* those with any contraindication to the technique proposed,

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-08 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
First analgesic request time | 24 hours post operatively
  The duration of effective analgesia is defined as the time from intrathecal injection to first patient analgesic demand

SECONDARY OUTCOMES:
Analgesic requirements | 24 hours post operatively
  A questionnaire will be used to record the analgesics consumed by the patients

CONTACTS AND LOCATIONS:
Overall Officials: Saleh Kanawati, MD, Principal Investigator — Makassed General Hospital
Locations (1):
- Makassed General Hospital, Beirut, Lebanon

REFERENCES:
- [Derived] Kanawati S, Barada MA, Naja Z, Rajab O, Sinno L, El Hasan J. Comparison of clinical effects of meperidine and sufentanil added to 0.5% hyperbaric bupivacaine for spinal anesthesia in patients undergoing cesarean delivery: a randomized controlled trial. J Anesth. 2022 Apr;36(2):201-209. doi: 10.1007/s00540-021-03031-6. Epub 2022 Jan 27. PMID 35083557